CLINICAL TRIAL: NCT01553513
Title: PET/CT for the Quantification of Atherosclerotic Plaque Inflammation in Patients With Coronary Heart Disease: The QAEK Trial
Brief Title: PET/CT for the Quantification of Atherosclerotic Plaque Inflammation
Acronym: QAEK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. med. M. Hacker, PD Dr. med. Marcus Hacker, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: PET; Coronary Artery Disease; Inflammation; Plaque; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Inflammation; Plaque, Amyloid; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 20 ml blood sample will be obtained from each patient. The following biomarkers will be assessed: glucose level, HBA1C, cholesterol levels, LDL cholesterol, HDL cholesterol, triglycerides, fibrinogen, factor XIII, plasminogen, complement C3, TNF-alpha, IL-6, CRP, resistin, adiponectin, CD40, 5-lipoxygenase, MMP-9, MMP-1, osteopontin, osteoprotegerin, fetuin, FGF21.
  ELISA and/or calorimetric assays will be used for the biochemical analyses of the serum markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1 - STEMI: Patients with acute cardiovascular event and typical aberrations in the ECG(STEMI) and positive serum markers
  Interventions: Other: [18F]-FDG positron emission computed tomography; Procedure: Invasive coronary angiography; Other: Serum biomarkers
- Group 2 - NSTEMI: Patients with acute coronary syndrome without typical aberrations in the ECG (NSTEMI) or without positive serum markers
  Interventions: Other: [18F]-FDG positron emission computed tomography; Procedure: Invasive coronary angiography; Procedure: Intravascular ultrasound and virtual histology; Other: Serum biomarkers
- Group 3 - symptomatic CAD: Symptomatic patients with stable CAD, who are eligible for ICA
  Interventions: Other: [18F]-FDG positron emission computed tomography; Procedure: Invasive coronary angiography; Procedure: Intravascular ultrasound and virtual histology; Other: Serum biomarkers
- Group 4 - STEMI: Patients eligible for ICA 6 months after STEMI and revascularization
  Interventions: Other: [18F]-FDG positron emission computed tomography; Procedure: Invasive coronary angiography; Procedure: Intravascular ultrasound and virtual histology; Other: Serum biomarkers

INTERVENTIONS:
Other: [18F]-FDG positron emission computed tomography — Patients will receive 20 mg furosemide and 20 mg butylscopolamine together with 370 MBq FDG. 120 minutes after the FDG application a ECG- and respiratory gated cardial PET acquisition will be performed, followed by a CT calcium scan, which will also be used for attenuation correction.
  This will be followed by CT-angiography with the application of 80 ml contrast medium. Patients without betablocker and a heart rate of more than 70 / min will be treated with 50 - 100 mg metoprolol as long as there are no contraindications.
  Subsequently, a 3D-mode whole body PET scan will be acquired followed by a low-dose CT transmission scan from the base of the scull to the iliac crest.
Procedure: Invasive coronary angiography — ICA is performed via the femoral artery in three projections (RAO 30°, RAO 15° and LAO 45°) and, if necessary, also in further projections. All angiograms are recorded digitally and assessed quantitatively by two experienced readers, who are blinded to the PET/CT results (Quant-Cor, QCA, Siemens Medical Systems, Forchheim, Germany or Digital Cardiac Imaging Systems, Philips, Eindhoven, Netherlands). The mean stenosis of the vessel is assessed in two projections and the percentage of stenosis is calculated for each single segment. Stenoses are localized by means of the AHA (American Heart Association) classification. Occlusions of the vessels are documented and revascularization is performed immediately in patients with acute coronary syndrome (STEMI, NSTEMI).
Procedure: Intravascular ultrasound and virtual histology — During the procedure an intravascular ultrasound will be recorded in grayscale. Radiofrequency raw-data will be collected at the peak of the R-wave and a VH-IVUS data recorder is used to reconstruct a color-coded map. Acquired data will be evaluated with a dedicated software. The grayscale IVUS images will be analyzed frame by frame and used to measure the diameter of the vessel lumen, of the external elastic membrane (EEM) as well as plaque and media thickness (defined as EEM minus lumen). The plaque burden will be calculated.
  A VH-IVUS analysis will be performed for each frame. Four plaque components will be color-coded: dense calcium white, the necrotic core red, fatty tissue light green and scar tissue dark green. color fractions are expressed as percentage of the plaque area and percentage of plaque volume.
  Lesions will be classified: pathologic intima thickening, fibroatheroma with thin cap, fibroatheroma with thick cap, fibrotic plaque and fibro-calcified plaque.
  Groups: Group 2 - NSTEMI; Group 3 - symptomatic CAD; Group 4 - STEMI
Other: Serum biomarkers — A 20 ml blood sample will be obtained from each patient. The following biomarkers will be assessed: glucose level, HBA1C, cholesterol levels, LDL cholesterol, HDL cholesterol, triglycerides, fibrinogen, factor XIII, plasminogen, complement C3, TNF-alpha, IL-6, CRP, resistin, adiponectin, CD40, 5-lipoxygenase, MMP-9, MMP-1, osteopontin, osteoprotegerin, fetuin, FGF21.
  ELISA and/or calorimetric assays will be used for the biochemical analyses of the serum markers.

SUMMARY:
This is a single-centre prospective trial with 140 patients employing [18F]-fluorodeoxyglucose positron emission computed tomography (FDG PET/CT) and advance motion correction and image fusion algorithms to create motion frozen displays and quantify FDG-uptake and thus inflammatory activity in atherosclerotic plaques in the coronary tree. Four groups of patients, two with stable coronary artery disease and two with acute coronary syndrome will be compared and the results of FDG PET/CT will be correlated to results of invasive coronary angiography, intravascular ultrasound / virtual histology, patient risk profile and serum markers of inflammation.

The investigators hypothesize that increased FDG accumulation in atherosclerotic plaques shows a positive correlation with inflammatory activity in coronary plaques and markers of plaque vulnerability as well as the risk profile of the patients and serum markers of inflammation. The investigators furthermore hypothesize that FDG PET/CT is able to detect high risk patients and provide an important means for risk stratification and optimization of patient management.

DETAILED DESCRIPTION:
Currently there are only morphological reference standards to detect vulnerable coronary plaques. However, inflammatory activity and plaque composition predict future cardiovascular events. Thus the aims and objectives of the study are the following:

1. Inflammatory activity of the coronary arteries and the great peripheral arteries shall be detected and quantified by means of FDG PET/CT hybrid imaging.
2. We aim to develop "motion frozen displays" of the heart and coronary arteries by means of ECG- and respiratory triggering of myocardial motion to reduce motion artifacts.
3. We aim to compare the coronary FDG uptake of patients with known stable CAD to the coronary FDG uptake of patients with acute coronary syndrome.
4. We aim to correlate coronary PET/CT with intravascular ultrasound (IVUS) / virtual histology (VH), which will be carried out during coronary angiography and provides the gold standard to characterize plaque composition.
5. Correlation of the inflammatory activity as measured by PET with the risk profile of the patients, blood coagulability and inflammatory and plaque-associated serum markers to establish a valid risk stratification.
6. Follow-up of the patients over at least one year to detect cardiovascular events.

Study Design

This is a prospective single-center study to evaluate coronary FDG PET/CT under controlled and standardized conditions. The study was approved by the local ethical committee as well as the German Federal Authority for Radiation Protection (Bundesamt für Strahlenschutz). All examinations will be performed at the University Hospital of the LMU in Munich. The study is in accordance with the Declaration of Helsinki, all patients provide informed written consent.

We plan to image four study populations with a high risk for inflammatory atherosclerosis or plaque rupture: two groups consist of patients with stable coronary disease and two groups consist of patients with acute coronary syndrome (Figure 1).

In the following, these groups will be described in more detail.

Patients with acute coronary syndrome Group 1: Patients with acute cardiovascular event and typical aberrations in the ECG (STEMI) and positive serum markers need to be stabilized immediately, thus they are not eligible for IVUS. However, by means of ICA the "culprit lesion" can be identified. 48 to 72 hours after the event the stable patients will receive FDG PET/CT to detect morphology and inflammation of the culprit lesion as well as further vulnerable plaques that might need intervention. PET/CT results will be correlated with results of ICA.

Group 2: Patients with acute coronary syndrome without typical aberrations in the ECG (NSTEMI) or without positive serum markers need to be stabilized immediately. In a second step ICA and IVUS / VH will be performed. 48 to 72 hours after the event the stable patients will receive FDG PET/CT to detect morphology and inflammation of the culprit lesion as well as further vulnerable plaques that might need intervention. PET/CT results will be correlated with results of ICA and IVUS / VH.

Patients with stable CAD Group 3: Symptomatic patients with stable CAD, who are eligible for ICA will receive and additional FDG PET/CT scan as well as IVUS / VH. Results will be correlated.

Group 4: Patients eligible for ICA 6 months after STEMI and revascularization will receive IVUS / VH and FDG PET/CT. Results will be correlated with regard to the former culprit lesion as well as further coronary lesions that might be present.

Summary of working hypotheses

Hypothesis 1 (technique) By means of FDG PET/CT the radiotracer uptake in the coronary arteries can be allocated to specific lesions and quantified with the aid of appropriate techniques for motion correction and three-dimensional image fusion.

Hypothesis 2 (association of FDG-uptake and extent of the disease) The coronary FDG-uptake of patients with stable CAD is significantly lower than the coronary FDG-uptake of patients with acute coronary syndrome.

Hypothesis 3 (correlation between IVUS/VH and FDG-uptake) Plaques with typical signs of vulnerability in IVUS/VH show a significantly increased FDG-uptake as a surrogate marker of inflammatory activity.

Hypothesis 4 (association of FDG-uptake and risk profile / serum markers) Coronary FDG-uptake shows a positive correlation with increasing risk profile (Framingham Score) and serum markers for plaque vulnerability and inflammatory reactions.

Hypothesis 5 (association of FDG-uptake and cardiovascular events) Increased coronary FDG-uptake and increased uptake in the peripheral vessels are associated with cardiovascular and cerebrovascular events over the course of one year.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients with known STEMI or NSTEMI and/or known CAD (see patient groups above)
* written informed consent for blood samples, ICA, IVUS/VH and FDG PET/CT

Exclusion Criteria:

* less than 50 years of age
* reason for symptoms other than coronary stenoses / occlusion
* known contraindication for the above listed examinations (like iodine allergy, intolerance of contrast media, claustrophobia)
* patients, who are not able to lie still without changing position over a minimum of 45 minutes
* pregnancy, breast feeding
* restricted renal function (creatinine > 1,5 mg% in women, > 2mg% in men)
* surgery within prior 24 hours

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary artery disease or with acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Association of FDG uptake and coronary plaque vulnerability | within 72 hours after enrollment
  Increased FDG uptake is found in plaques that fulfill the criteria of plaque vulnerability as measured with IVUS/VH.

SECONDARY OUTCOMES:
Association of FDG-uptake and extent of the disease | within 72 hours after enrollment
  The coronary FDG-uptake of patients with stable CAD is significantly lower than the coronary FDG-uptake of patients with acute coronary syndrome.
Association of FDG-uptake and risk profile / serum markers | within 72 hours after enrollment
  Coronary FDG-uptake shows a positive correlation with increasing risk profile(Framingham Score) and serum markers for plaque vulnerability and inflammatory reactions.
Association of FDG-uptake and cardiovascular events | within 1 year of follow-up
  Increased coronary FDG-uptake and increased uptake in the peripherial vessels are associated with cardiovascular and cerebrovascular events over the course of one year.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hacker, MD, Principal Investigator — LMU Munich
Locations (1):
- Department of Nuclear Medicine, Departmen of Cardiology, University of Munich, Munich, Bavaria, Germany